CLINICAL TRIAL: NCT06224647
Title: Effectiveness and Uptake of a Transdiagnostic Emotion Regulation Mobile Intervention Among University Students: A Randomized Controlled Trial
Brief Title: Evaluation of a Transdiagnostic Mobile App Intervention Among University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus University Rotterdam (Other)
Responsible Party: Principal Investigator, Marilisa Boffo, Assistant professor of Clinical Psychology and eHealth, Erasmus University Rotterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ETH2324-0193
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Emotion Regulation; Stress; Resilience; Depressive Symptoms; Anxiety
Keywords: Transdiagnostic intervention; Digital intervention; Mental health; University Students; Randomized Controlled Trial
MeSH Terms: conditions — Emotional Regulation; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study is a 12-week superiority parallel-group randomized controlled trial including three follow-up assessments at weeks 3, 8, and 12. Eligible participants are randomized to either an intervention condition (i.e., full access to the app) or to the waitlist control condition (i.e., receives access upon completion of the study).
Who Masked: Investigator
Masking Description: The investigator conducting the analyses will be blinded to group assignments, remaining unaware of which data corresponds to the control group and which to the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to the intervention (Experimental): Participants assigned to the intervention group will have full access to the mobile app intervention, namely ROOM app, for the whole duration of the 12-week trial.
  As part of the app's onboarding process, participants will receive tips on optimal app usage and can decide to take part in a 21-day challenge where they are encouraged to assess their emotional states on a daily basis and complete one exercise per day. During the onboarding process, participants are encouraged to explore different emotional regulation exercises offered in the app and to save the ones they find most beneficial in their "virtual Room", curating a personalized well-being toolkit. While daily notifications prompt regular app engagement, no additional efforts are made to further promote its use.
  Interventions: Behavioral: Mobile Transdiagnostic Emotion Regulation Intervention
- Waitlist control condition (No Intervention): Participants allocated to the control group will be put on a waitlist and granted access to the mobile intervention after the trial concludes. They will then receive the same intervention with the identical onboarding process as the intervention group.

INTERVENTIONS:
Behavioral: Mobile Transdiagnostic Emotion Regulation Intervention — The intervention aims to provide a tailored and engaging way for users to manage and comprehend their emotional well-being.
  It consist of 5 components:
  1. Daily tracking of emotions
  2. A suite of exercises placed in six categories facilitating adaptive emotion regulation skills (i.e., upregulation of positive effect, self-compassion, cognitive defusion and cognitive restructuring, mindfulness, breathing techniques),
  3. A self-assessment module where users can complete surveys evaluating their states (e.g., wellbeing) and traits (e.g., perfectionistic tendencies),
  4. A personal toolkit area (i.e., each exercise is represented by an object commonly found in a student's room. Users can collect objects of favoured exercises in the virtual ROOM, enabling them quick access to exercises they liked / found helpful),
  5. A recommendation system linking users to the content based on their specific needs or preferences
  Other Names: ROOM app
  Arms: Access to the intervention

SUMMARY:
This study is a two-armed randomized controlled trial (RCT) aimed at evaluating the effectiveness and adoption of a transdiagnostic mobile app intervention that focuses is on enhancing adaptive emotional regulation (ER) skills among university students.

DETAILED DESCRIPTION:
Globally, an estimated 30% of university students struggle with mental health issues, primarily anxiety, depression, and substance abuse. Recent trends have highlighted the potential of online interventions for accessible, low-threshold support in preventing these issues among this demographic.

At Erasmus University Rotterdam (EUR), a transdiagnostic mobile app is being developed as part of a student wellbeing program. This app provides a range of tools aimed at improving mental health by teaching students adaptive emotional regulation strategies. It incorporates exercises from various therapeutic modalities, addressing factors like negative thoughts, rumination, and prolonged negative emotions. Delivered through a smartphone, the app includes 24 therapeutic exercises focusing on techniques such as enhancing positive emotions, mindfulness, cognitive defusion, cognitive restructuring, relaxation, breathing, and self-compassion.

The present study is a 12-week two-armed RCT study with outcomes assessed at the baseline, and three follow-ups at weeks 3, 8, and 12. It compares a group of distressed students with access to the mobile app intervention against a waitlist control group.

The main goal of the study is to assess the impact of the intervention on stress symptoms and emotional regulation skills. The secondary outcomes of the study, include an evaluation of the intervention's impact on depression, anxiety symptoms, and students' resilience levels. Lastly, the study examines the app's uptake, including engagement patterns and user experiences, and evaluates the real-life application of the skills learned through the app.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate and provide informed consent
* Access to smartphone and internet
* Feels comfortable with English language for verbal and written communication and interaction with the app
* Scores <13 on the Perceived Stress Scale (PSS-10)

Exclusion Criteria:

* Scores >20 on the Patient Health Questionnaire (PHQ-9)
* Having a medical diagnosis of psychosis or bipolar disorder, severe clinical depression or anxiety disorder
* Undergoing psychopharmacological treatment or treatment with experimental drugs

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in stress symptoms | At baseline and days 21, 56, and 84.
  Perceived Stress Scale (PSS-10) is used to evaluate participants' stress levels. Participants are asked to specify how often they felt or thought a certain way over the last month on a scale from 0 [never] to 5 [very often]. The score ranges from 0 - 40, with higher scores indicating higher levels of perceived stress symptoms.
Changes in ER skills | At baseline, and days 56 and 84.
  The Emotion Regulation Skills Questionnaire (ERSQ) will be used to assess emotion regulation skills. This instrument includes seven distinct emotion regulation skills: awareness, sensation, clarity, understanding, acceptance, tolerance, compassionate self-support, confrontation readiness, and modification of negative emotions. It consists of 27 items, each scored on a scale ranging from 0 (not at all) to 4 (almost always). Higher scores on both the ERSQ subscales and the aggregate ERSQ score are indicative of higher emotion regulation skills.

SECONDARY OUTCOMES:
Changes in depressive symptoms | At baseline and day 84
  Depressive symptoms are measured with the Patient Health Questionnaire (PHQ-9). Participants are asked to indicate how often they have been bothered by a certain symptom over the past two weeks on a scale from 0 (not at all) to 3 (nearly every day). PHQ-9 scores range from 0-27. Higher scores indicate higher levels of depressive symptoms.
Changes in anxiety symptoms | At baseline and day 84
  Anxiety symptoms are measured with the Generalized Anxiety Disorder (GAD-7) questionnaire. Participants are asked to indicate how often they have been bothered by a certain symptom over the last two weeks on a scale from 0 (not at all) to 3 (nearly every day). The scores on GAD-7 range between 0-21, with higher scores indicating higher levels of anxiety.
Changes in resilience levels | At baseline and day 84
  Resilience levels are evaluated with the 10-item Connor-Davidson Resilience Scale (CD-RISC-10). Items are scored on a scale ranging from 0 (not true at all) to 4 (true nearly all the time). Total scores range between 0 and 40 with higher scores indicating greater resilience.
Objective engagement patterns | Day 1 - 84
  Objective engagement patterns include exercise completion and non-completion (i.e., exercise started but not finished) rates, average time spent on each exercise, engagement in self-assessment module (i.e., number of questionnaires and Ecological Momentary Assessments completed), the number of objects collected in the "virtual room", the number of times the app was accessed. Log data is used to evaluate objective engagement patterns.
Subjective engagement: Exercise likeability and helpfulness | Day 1-84
  Exercise likeability and helpfulness is evaluated on a 5-point Likert scale ranging from 1 (not at all) to 5 (very much) every time a participant completes an exercise.
  * How much did you like the exercise?
  * How helpful did you find the exercise?
Subjective engagement: Likeability and helpfulness of Self-assessment component | Day 56
  The likeability and helpfulness of the Self-assessment module (MapMyself) is evaluated on a scale from 1 (not at all) to 5 (very much)
  * How much did you like the self-assessment (MapMyself) feature in the app?
  * How helpful did you find the self-assessment (MapMyself) feature in the app?
Subjective engagement: Likeabilty of Virtual Collectibles Room | Day 56
  The likeability of the Virtual Collectibles Room component is assessed on a scale ranging from 1 (not at all) to 5 (very much)
  - How much do you like collecting objects in the ROOM app?
Subjective engagement: Usefulness and perceived effectiveness of recommendation system | Day 56
  Participants are asked to evaluate the recommendation system by rating the following two questions on a scale from 1 (not at all) to 5 (very much)
  * How useful do you find the in-app recommendations of the exercises?
  * How well do the in-app recommendations of exercises align with your self-reported moods?
Subjective engagement: User experience with the app | Day 56
  User experiences are evaluated with a User Experience Questionnaire (UEQ) measuring the Attractiveness, Perspicuity, Efficiency, Dependability, and Novelty of the app. The questionnaire includes 26 items measured on a semantic differential (e.g., attractive - unattractive). The items are scored from -3 (the most negative answer) to +3 (the most positive answer), with 0 representing a neutral answer.
Engagement with the exercises outside of the app: In app counter | Day 1-84
  The mobile intervention includes a feature (i.e., an exercise counter) where users can log in the number of times they completed an exercise outside of the app.
  This counter is used to evaluate the number of exercises performed independently from the app.
Engagement with ER techniques outside of the app | Day 21, 56, 84
  Participants are asked to evaluate how often they applied ER techniques (e.g., self-compassion, breathing pattern, savouring, being mindful, reframing unhelpful thoughts) in their daily life over the past month on a scale from 0 (not at all) - 4 (daily).
  - Over the past month, how frequently have you spontaneously used any of the techniques you've learned in ROOM app either to manage your emotions during challenging times or to improve your overall mood?
Likability and helpfulness of transfer strategies offered in the app | Day 56
  For evaluation of the learning transfer features in the app, participant will be asked to rate the following questions on a scale from (0 - Not at all; 100 - Very much or So far I haven't used this feature).
  * How much do you like action planning with 'when-then' statements?
  * How helpful do you find the action planning with 'when-then' statements?
  * How much do you like to use stickers to create cues to practice the techniques?
  * How helpful do you find stickers to create cues to practice the techniques?
  * How much do you like the 'practice semi-guided' feature of the app?
  * How helpful do you find the 'practice semi-guided' feature of the app?

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus University Rotterdam, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data [and code] produced in the project will be shared in a research data repository [EUR Data Repository (EDR) and Open Science Framework (OSF)]. A DCMI (Dublin Core Metadata Initiative) standard will be used to document this research. There will be a temporary restriction on re-using of the data (Embargo period of 6 months).
  Data (and code) that will be shared in a research data repository are: Anonymized survey data, Codebook and Blank Questionnaires, Readme text file (general description of the data, including date of collection, selection procedure of participants, tools used to collect the data etc.), and scripts of data analysis.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data will come available after the embargo period of 6 months

REFERENCES:
- [Background] Laure T, Engels RCME, Remmerswaal D, Spruijt-Metz D, Konigorski S, Boffo M. Optimization of a Transdiagnostic Mobile Emotion Regulation Intervention for University Students: Protocol for a Microrandomized Trial. JMIR Res Protoc. 2023 Oct 27;12:e46603. doi: 10.2196/46603. PMID 37889525